CLINICAL TRIAL: NCT04553497
Title: Does Interferential Current Provide Additional Benefit to the Rehabilitation Program for the Patients With Proximal Humeral Fractures? A Randomized Controlled Study
Brief Title: IFC Therapy in Proximal Humerus Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Emine Duran, Medical doctor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-10.1/43
Record Dates: First submitted 2020-09-08; First posted 2020-09-17 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Interferential Current in Proximal Humerus Fractures
Keywords: Proximal humerus fracture; interferential current; Constant-Murley score
MeSH Terms: interventions — Electric Stimulation Therapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: After the patients were randomized, interferential current was applied for 3 times a week before the each exercise session by another physiotherapist. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. Subjects were told that in order to produce an effect, the intensity of the stimulator must be maintained at a "strong but comfortable level" at all times. The sham interferential current therapy consisted of the placement of the same pads for the same time but no electrical stimulation was applied to the probes.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients and the outcome assessor were blind to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation and interferential current therapy (Active Comparator): Flipping a coin was used for simple randomization (tails - interferential current). In this arm, interferential current therapy was applied to the patients in addition to the rehabilitation program.
  Interventions: Device: Interferential current; Other: Rehabilitation program
- Rehabilitation and sham therapy (Sham Comparator): Flipping a coin was used for simple randomization (heads - sham). In this arm, sham therapy was applied to the patients in addition to the rehabilitation program.
  Interventions: Device: Interferential current; Other: Rehabilitation program

INTERVENTIONS:
Device: Interferential current — Interferential current or sham were applied to the patients before the each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. Subjects were told that in order to produce an effect, the intensity of the stimulator must be maintained at a "strong but comfortable level" at all times. The sham interferential current therapy consisted of the placement of the same pads for the same time but no electrical stimulation was applied to the probes.
Other: Rehabilitation program — The orthopedic rehabilitation programme was applied to all patients three times a week for 4 weeks under the guidance of the same physiotherapist. The first phase (0-3 weeks) involved the elbow, wrist, and hand active range of motion (ROM) and pendulum (clockwise and counterclockwise) exercises in the 0-2 weeks of the non-displaced fracture. For displaced fractures, elbow, wrist, and hand active range of motion was started immediately, but pendulum exercises were initiated two weeks later. The patients were instructed to continue exercises 3-5 times per day for 30 minutes. After two weeks, active assistive ROM and isometric exercises were performed supine position. During the second phase (3-6 weeks), active forward elevation in supine was carried out and then progressed to sitting and standing position. At the end of the sixth week, a home exercise program was given by the physiotherapist, including resistance exercises using an elastic band (Thera-Band).

SUMMARY:
Proximal humerus fractures (PHFs) frequently occur in the elderly and osteoporotic population, but these fractures are also common in individuals under age 60 years. Conservative treatment of PHF usually involves a short period of immobilization followed by orthopedic rehabilitation. However, the severe pain of some patients with fractures limits their participation in the exercise programme, and shoulder muscle atrophy and frozen shoulder may occur in these patients due to immobilization. There are conflicting results regarding the use of physical therapy modalities in the shoulder pain management. Interferential current (IFC) therapy is believed to be effective for the pain-relieving through several mechanisms. Although IFC has been investigated in many painful shoulder disorders, there is no reported study on the effectiveness of IFC therapy in patients with PHF. This study aimed to investigate the effectiveness of IFC added to exercise on shoulder function, pain, and disability compared with placebo in patients with conservative treated PHF.

Patients were evaluated within the first week of PHF and divided into two groups to receive either IFC or sham using a simple randomization method. The orthopedic rehabilitation programme was applied to all patients three times a week for four weeks under the guidance of the same physiotherapist. IFC or sham therapy was applied three times a week for 20 minutes before each exercise session by another physiotherapist.

Shoulder functions, pain (visual analogue scale), disability and range of motion was evaluated at the end of the rehabilitation program, at 6-weeks and 18-weeks post-treatment by the physiatrist (ED) who did not know which group the patients belonged to. In addition, the amount of acetaminophen usage was noted at each visit.

DETAILED DESCRIPTION:
Patients with conservatively treated proximal humerus fracture who admitted to Ege University Physical Medicine and Rehabilitation outpatient clinic have been included in the study. All patients who met inclusion criteria were enrolled into the study at the first week of PHF. The orthopedic rehabilitation programme was applied to all patients three times a week for four weeks under the guidance of the same physiotherapist. The patients also received a complete set of premade exercise cards, which showed all exercises to ensure that the training program was learned correctly. The patients were recruited at the first week after proximal humerus fracture and then allocated into the groups. The patients were separated into two groups as interferential current or sham using a simple randomization method managed by an impartial observer. Flipping a coin was used for simple randomization (heads - sham, tails - treatment). The patient's group was reported to the physiotherapist who would apply interferential current in a closed envelope. Patients and the outcome assessor were blind to the treatment groups. The IFC therapy was applied using a combined electrotherapy device SONOPULS 692® (brand: Enraf-Nonius). The medium frequency of the IFC was 4000 Hz and 4100 Hz to produce the amplitude-modulated frequency at 100 Hz. Two rubber electrodes (8×6 cm) were fitted on the fractured shoulder. One of the electrodes was placed on the lateral part of the deltoid muscle; the other one was placed on the trapezius muscle near the shoulder. The current intensity was set to achieve a "strong but comfortable tingling" without visible muscle contraction. The sham therapy consisted of placing the same pads for the same time, but no electrical stimulation was applied to the probes. The primary outcome was shoulder global function which was measured by the Constant-Murley score (CMS). The questionnaire assesses four shoulder functions: 1) pain; 2) activities of daily living (sleeping, work, leisure); 3) range of motion; and 4) muscle strength. The total score ranges from 0 to 100, with a higher score indicating better shoulder function. Activity pain was measured with the visual analog scale (VAS). In addition, in order to evaluate shoulder function and disability, the Disability of the Arm, Shoulder and Hand questionnaire (DASH) was used. This self-administered questionnaire includes 30 questions evaluated on a 5-point Likert scale, most of which relate to the individual's capacity to realize a task. The patients were allowed to use paracetamol during the study and the paracetamol intake was recorded as gr/week.

Clinical assessments were evaluated at the end of the treatment, at 6-weeks and 18-weeks post-treatment. Only VAS resting pain was evaluated at the enrollment because the fractured side was immobile when the patients were included in the study. The physician who assessed the treatment outcomes, the patients and the physiotherapist who administer the exercises were unaware of the patient's group of treatment.

A clinically meaningful difference was considered to be a change of 15 points in total CMS. In order to detect this improvement, the number of patients needed was 17 per group according to a power of 0.80, a high size effect (d=0.88), a p value of 0.05, and a 15% dropout rate.

Statistical analysis was performed using SPSS version 20.0 (IBM, Armonk, NY, USA). An intention-to-treat analysis was employed for all analysis. The variables were investigated using visual (histogram, probability plots) and analytic methods (Kolmogorov-Smirnov, skewness and curtosis) to determine whether they were normally distributed or not. . Continuous data were described as median (inter-quartile range, IQR) or mean (standar deviation, SD) and categorical variables as percentages. Chi-square or Fisher's exact test was used to compare categorical variables and Mann-Whitney U test/Student's T-test was used to compare continuous variables. All outcome values were presented in mean and standard deviation. The repeated measures ANOVA test was used in comparison of the means of the repeated measures. The results of the repeated measures ANOVA were analyzed by Mauchly's sphericity test. If the parametric tests (factorial design for repeated measures analysis) did not provide the preconditions, the Greenhouse-Geisser correction was used for corrections to the degrees of freedom or Friedman's Test. The Bonferroni correction was used for multiple comparisons. A p value of less than 0.05 was considered to show a statistically significant result.

ELIGIBILITY:
Inclusion criteria were as follows: age ≥ 40 years, PHFs did not require surgery by the orthopedic surgeon, and admission to our outpatient clinic within the first two weeks after the fracture

Exclusion Criteria:

* Any surgery history for shoulder pathologies
* Previous electrotherapy experience before the fracture (to ensure blinding of therapy)
* Any contraindication such as pacemaker, malignancy, pregnancy, etc. for IFC
* Rheumatic disease such as rheumatoid arthritis and ankylosing spondylitis
* Shoulder subluxation; having other fractures in addition to the PHF
* Known or suspected joint infection or a specific condition such as peripheral or central nervous system lesions
* Neoplasm; diabetes mellitus or osteonecrosis
* Any mental disorder that may make it difficult to adapt to exercise

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emine Duran, Principal Investigator — Ege University, School of Medicine, Physical Medicine and Rehabilitation; Berrin Durmaz, Study Director — Ege University, School of Medicine, Physical Medicine and Rehabilitation; Funda A Çalış, Study Chair — Ege University, School of Medicine, Physical Medicine and Rehabilitation; Mehmet R Kadı, Study Chair — Ege University, School of Medicine, Physical Medicine and Rehabilitation; Levent Küçük, Study Chair — Ege University, School of Medicine, Orthopaedic Surgery
Locations (1):
- Ege University, School of Medicine, Department of Physical Medicine and Rehabilitation Outpatient Clinic, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodgson SA, Mawson SJ, Stanley D. Rehabilitation after two-part fractures of the neck of the humerus. J Bone Joint Surg Br. 2003 Apr;85(3):419-22. doi: 10.1302/0301-620x.85b3.13458. PMID 12729121
- [Result] Hodgson S. Proximal humerus fracture rehabilitation. Clin Orthop Relat Res. 2006 Jan;442:131-8. PMID 16394751
- [Result] Cheing GL, So EM, Chao CY. Effectiveness of electroacupuncture and interferential eloctrotherapy in the management of frozen shoulder. J Rehabil Med. 2008 Mar;40(3):166-70. doi: 10.2340/16501977-0142. PMID 18292916
- [Result] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 who met the study inclusion criteria were randomly separated into two groups: the interferential current group (n = 18) and the sham group (n =17).
Pre-assignment Details: 18 patients were excluded
  * Rheumatic diseases, 6
  * Multiple trauma, 5
  * Cerebrovasculer diseases, 3
  * Peripheral nerve injury, 2
  * Shoulder subluxation, 2
Groups:
- Rehabilitation and Sham Therapy: Flipping a coin was used for simple randomization (heads - sham). In this arm, sahm interferential current therapy was applied to the patients in addition to the rehabilitation program.
  Sham interferential current was applied to the patients before each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. The sham interferential current therapy consisted of the placement but no electrical stimulation was applied to the probes. Rehabilitation program was performed to all patients.
- Rehabilitation and Interferential Current Therapy: Flipping a coin was used for simple randomization (tails - interferential current). In this arm, interferential current therapy was applied to the patients in addition to the rehabilitation program.
  Interferential current: Interferential current was applied to the patients before each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. Subjects were told that in order to produce an effect, the intensity of the stimulator must be maintained at a "strong but comfortable level" at all times.
  Rehabilitation program was performed to all patients
Period: Overall Study
Arm/Group | Rehabilitation and Sham Therapy | Rehabilitation and Interferential Current Therapy
Started | 17 | 18
Completed | 15 | 17
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Rehabilitation and Interferential Current Therapy: In this arm, interferential current therapy was applied to the patients in addition to the rehabilitation program. Interferential current: were applied to the patients before the each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. Subjects were told that in order to produce an effect, the intensity of the stimulator must be maintained at a "strong but comfortable level" at all times.
  Rehabilitation program: Rehabilitation program carried out under the guidance of same physiotherapist 3 times a week for 6 weeks. At the end of 6 weeks', the physiotherapist described the home training program involving the resistance exercises by using therabands
- Rehabilitation and Sham Therapy: In this arm, sham interferential current therapy was applied to the patients in addition to the rehabilitation program.
  Sham interferential current were applied to the patients before the each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. The sham interferential current therapy consisted of the placement of the same pads for the same time but no electrical stimulation was applied to the probes.
  Rehabilitation program: Rehabilitation program carried out under the guidance of same physiotherapist 3 times a week for 6 weeks. At the end of 6 weeks', the physiotherapist described the home training program involving the resistance exercises by using therabands.
- Total: Total of all reporting groups
Arm/Group | Rehabilitation and Interferential Current Therapy | Rehabilitation and Sham Therapy | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.7) | 62.0 (9.5) | 60.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Turkey | 18 | 17 | 35
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (3.2) | 30.8 (5.6) | 29.3 (4.7)
Fracture side [Count of Participants; unit: Participants]
  Right fracture | 15 | 15 | 30
  Left fracture | 3 | 2 | 5
Neer classification [Count of Participants; unit: Participants] — The Neer classification divides the proximal humerus into four parts and considers not the fracture line, but the displacement as being significant in terms of classification. The four parts are the humeral head, the greater tuberosity, the lesser tuberosity and the humeral shaft. Displacement is on a per-part basis. Minimal displaced fractures are named as Neer Type-1. Fractures involving> 1 cm or 45° angular displacement are named as Neer Type-2, Type-3 and Type-4 according to the number of displaced fracture parts.
  Participants
    Type-1 Neer Classification | 4 | 2 | 6
    Type-2 Neer Classification | 3 | 6 | 9
    Type-3 Neer Classification | 11 | 9 | 20
Anatomic segment of proximal humerus fracture [Count of Participants; unit: Participants] — The anatomical part of the proximal humerus fracture is divided into four parts as anatomical neck, surgical neck, lesser tuberosity, and greater tuberosity.
  Participants
    Greater tuberosity fracture | 5 | 3 | 8
    Surgical neck fracture | 2 | 5 | 7
    Greater tuberosity and Surgical neck fracture | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Constant-Murley Score
Description: The primary outcome was shoulder global function which was measured by the Constant-Murley score (CMS). The questionnaire assesses four shoulder functions: 1) pain; 2) activities of daily living (sleeping, work, leisure); 3) range of motion; and 4) muscle strength. The total score ranges from 0 to 100, with a higher score indicating better shoulder function.
Time Frame: 1. At the end of the treatment 2. The second evaluation: Six weeks after the first one (6th week post-treatment) 3. The last evaluation: Three months after the second one (18th week post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rehabilitation and Interferential Current Therapy: In this arm, interferential current therapy was applied to the patients in addition to the rehabilitation program.
- Rehabilitation and Sham Therapy: Sham therapy was applied to the patients in addition to the rehabilitation program.
Arm/Group | Rehabilitation and Interferential Current Therapy | Rehabilitation and Sham Therapy
Number analyzed (Participants) | 18 | 17
score on a scale
  Post treatment (Constant-Murley scores) | 57.0 (7.7) | 48.2 (12.0)
  6th week post-treatment (Constant-Murley scores) | 69.0 (8.9) | 60.7 (12.1)
  18th week post-treatment (Constant-Murley scores) | 79.6 (9.4) | 69.3 (14.2)

2. Secondary Outcome: Visual Analogue Scale
Description: The secondary outcome was pain which was measured by the visual analogue scale. The patients themselves used the VAS to make an assessment of their pain with 0 representing no pain, 10 cm representing severe pain.
Time Frame: Visual analogue scale was recorded at the end of the treatment, at 6-weeks and 18-weeks post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rehabilitation and Sham Therapy: Sham interferential current therapy was applied to the patients in addition to the rehabilitation program.
Arm/Group | Rehabilitation and Interferential Current Therapy | Rehabilitation and Sham Therapy
Number analyzed (Participants) | 18 | 17
score on a scale
  VAS at the post-treatment | 3.9 (1.5) | 4.7 (1.5)
  VAS at 6-weeks post-treatment | 2.0 (1.7) | 3.0 (1.5)
  VAS at 18-weeks post-treatment | 0.7 (1.1) | 1.7 (1.4)

3. Secondary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH) Score
Description: One of the secondary outcome was disability which was measured by the Disabilities of the Arm, Shoulder and Hand (DASH) Score. The DASH consists mainly of a 30-item disability/symptom on a 5-point Likert scale, scored 0 (no disability) to 100 (maximum disability).
Time Frame: Disabilities of the Arm, Shoulder and Hand (DASH) Score was recorded at the end of the treatment, at 6-weeks and 18-weeks post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rehabilitation and Interferential Current Therapy | Rehabilitation and Sham Therapy
Number analyzed (Participants) | 18 | 17
score on a scale
  DASH score at post-treatment | 28 (11) | 38.4 (17.5)
  DASH score at 6-weeks post-treatment | 15.3 (9.2) | 23.3 (13)
  DASH score at 18-weeks post-treatment | 7.7 (7.3) | 12.5 (11.3)

ADVERSE EVENTS:
Time Frame: For 22 weeks after the fracture
Groups:
- Rehabilitation and Interferential Current Therapy: In this arm, interferential current therapy was applied to the patients in addition to the rehabilitation program.
  Interferential current was applied to the patients before the each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. One electrode was placed on the lateral part of the deltoid muscle; the other was placed on the trapezium muscle close to the shoulder. Subjects were told that in order to produce an effect, the intensity of the stimulator must be maintained at a "strong but comfortable level" at all times.
  Rehabilitation program carried out under the guidance of same physiotherapist 3 times a week for 6 weeks. At the end of 6 weeks', the physiotherapist described the home training program involving the resistance exercises by using therabands.
- Rehabilitation and Sham Interferential Current Therapy: Sham interferential current therapy was applied to the patients in addition to the rehabilitation program.
  Sham interferential current was applied to the patients before the each exercise session. Pre-modulated bipolar method with the currier frequency of 4 kHz by a combination therapy unit (Sonopuls 692, Enraf-Nonius) with two electrodes (8×6 cm) was used. The sham interferential current therapy consisted of the placement of the same pads for the same time but no electrical stimulation was applied to the probes.
  Rehabilitation program carried out under the guidance of same physiotherapist 3 times a week for 6 weeks. At the end of 6 weeks', the physiotherapist described the home training program involving the resistance exercises by using therabands.
Arm/Group | Rehabilitation and Interferential Current Therapy | Rehabilitation and Sham Interferential Current Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No